CLINICAL TRIAL: NCT06502639
Title: Effects of Tharaplay Program on Hand Dexterity in Children With Hemiplegic Cerebral Palsy
Brief Title: Effects of Theraplay on Hand in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0777
Record Dates: First submitted 2024-06-11; First posted 2024-07-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: cp; hand dexterity; theraplay

STUDY DESIGN:
Intervention Model Description: it will randomized controlled trial in which non probability convenient sampling will be used. Two groups of 6-12 years will be performed in which participant will randomly divided. Group A will recieve conventional therapy and Group B will recieve conventional therapy with theraplay program.
Who Masked: Participant
Masking Description: participant will get seperate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional therapy (Active Comparator): The control group will receive a designed conventional physical therapy program for the affected hand like stretching and strengthening exercises, sponge ball exercises to the hand, and hand weight bearing exercises.
  Interventions: Other: conventional physical therapy
- conventional therapy along with theraplay program (Experimental): The experimental group will receive Theraplay therapy or a program and different play-based activities like playing with wooden puzzles and playing with clay and blocks, special handshake claps high fives, making wraps, and bubble tennis in addition to designed conventional therapy.
  Interventions: Other: theraplay program

INTERVENTIONS:
Other: theraplay program — A play therapy method called "thermaplay" aids in children's development of stronger bonds and relationships with others. It emphasizes the parts of communication that are nonverbal. When it comes to giving cerebral palsy children with hand therapy that is both effective and motivating, fun approaches have been shown to be both successful and appealing.
  Arms: conventional therapy along with theraplay program
Other: conventional physical therapy — conventional physical therapy program for like stretching and strengthening exercises, sponge ball exercises to the hand, and hand weight bearing exercises
  Arms: conventional therapy

SUMMARY:
Among the neurological conditions known as cerebral palsy are those that impact muscle tone, mobility, and cooperation. Cerebral palsy that affects only one side of the body is known as hemiplegic cerebral palsy. Damage to one side of the brain causes this disorder, which usually manifests as before, in the middle of, or soon after birth. The ability to use one's hands with coordination and expertise to accomplish tasks that call for control and accuracy is known as hand dexterity. For those who have cerebral palsy, hand dexterity can be a major issue. Developing hand dexterity is crucial as it might augment an individual's capacity to execute routine tasks and attain greater autonomy.Convenient sampling will be used to carry out a randomized control study.

Twenty two subjects will be divided into two groups at random. The experimental group will receive Theraplay therapy, which is a program that includes various play-based activities like playing with wooden puzzles, clay and blocks, making wraps, bubble tennis, and special handshakes, claps, and high fives, in addition to designed conventional therapy. The control group will receive designed conventional physical therapy exercises for the affected hand, such as hand weight-bearing exercises, stretching and strengthening exercises, and exercises using sponge balls.

The course of treatment will run for eight weeks. As outcome measures, the GMFCS and MACS scales, the box and block test, finger tapping, and the nine-hole peg test will be employed.

Data will be analyzed on SPSS version 25; the normality of the data will be checked and tests will be applied according to the normality of the data either it will be a parametric test or non parametric based on the normality.

DETAILED DESCRIPTION:
Group A: The control group will receive a designed conventional physical therapy program for the affected hand like stretching and strengthening exercises, sponge ball exercises to the hand, and hand weight bearing exercises.

Group B: The experimental group will receive Theraplay therapy or a program and different play-based activities like playing with wooden puzzles and playing with clay and blocks, special handshake claps high fives, making wraps, and bubble tennis in addition to designed conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ages of both boys and girls range from 6 to 12 years
* Based on the Modified Ashworth Scale, the degree of spasticity is between 1 and 1+.
* Capable of grasping, releasing, and reaching with the afflicted hand
* Capable of comprehending and adhering to instructions

Exclusion Criteria:

* Children with mixed C.P., ataxic, athetoid, and mental retardation
* Visual and auditory issues
* Upper limb congenital malformations, Convulsions
* Youngsters who have recently sustained upper extremity trauma

Ages: 6 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
modified ashworth scale | 8 weeks
  The Modified Ashworth Scale (MAS) is a commonly used clinical assessment tool to evaluate muscle tone and spasticity in individuals with neurological conditions such as spastic cerebral palsy. It is a reliable and valid method for grading muscle resistance during passive movement. interrater reliability of AS and MAS varied from moderate to good. ICC scores of AS were between 0.54 and 0.78 and MAS were between 0.61-0.87. Test-retest results of AS and MAS varied from poor to good. ICC values were between 0.31 and 0.82 for AS and between 0.36 and 0.83 for MAS.
ABILHAND-KID | 8 Weeks
  a clinical instrument for assessing children with cerebral palsy's physical dexterity. The parents rated 21 largely bimanual elements that made up the ABILHAND-Kids scale. Because the parents gave a more accurate assessment of their kids' abilities than the kids did, the measurement range was larger, the reliability (R=0.94) was higher, and the results were consistent over time.
Manual Ability Classification scale | 8 weeks
  The purpose of the Manual Ability Classification System is to categorize the ways in which kids with cerebral palsy use their hands to handle items during everyday tasks. The categorization is intended to represent the child's average manual performance rather than their maximum ability. There are five levels to it.
Gross Motor Functional Classification Scale | 8 weeks
  The most widely used scale by pediatric professionals to characterize the degree of gross motor impairment in children with cerebral palsy is the GMFCS. The five-level Gross Motor Function Classification System is used to categorize children with cerebral palsy according to their current gross motor ability, their limits in gross motor function, and whether or not they require assistive technology or wheeled mobility.
Box And Block Test | 8 weeks
  During therapy, a functional test called the Box and Blocks Test is performed to gauge a child with cerebral palsy's gross manual dexterity. The exam consists of a box with a center partition.
Nine Hole Peg Test | 8 weeks
  Patients with cerebral palsy can have their finger dexterity measured with the Nine Hole Peg Test.The patient picks up each of the nine pegs as fast as they can and inserts them into the nine holes in this test using a start command that starts a stopwatch.
Finger Tapping Test | 8 weeks
  The Finger Tapping Test, sometimes called the Tapping Speed Assessment, is one of the many tools available to assess motor control and the condition of the neuromuscular system.

CONTACTS AND LOCATIONS:
Overall Officials: sidra jamal, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Tahsin Z. Effect of hand activities group therapy program on ADL performance of children with cerebral palsy at CENTRE FOR THE REHABILITATION OF THE PARALYSED (CRP): Bangladesh Health Professions Institute, Faculty of Medicine, the University …; 2019.